CLINICAL TRIAL: NCT04864301
Title: Tumescent Stretching Measurment Technique: A New Technique for Intraoperartive Measurement of Inflatable Penile Implant Size
Brief Title: Tumescent Stretching Measurement Technique
Acronym: TSMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adham ZAAZAA, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSMT
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: To Try to Eliminate Frequencies of Insertions in Order to Arrive to Adequate Size of Implanted Penile Prosthesis
Keywords: penile implant, iflatable penile implant, re-insertion, measurement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tumescent Stretching Measurement Technique (Active Comparator): The "Tumescent Stretching Measurement Technique" (TSMT) group (N=12) will be administered an intracorporal injection (ICI) of 20 microgram Alprostadil. Hegar 7 dilator will be introduced through the corporotomy until reaching a bone stopping point. The tumescent penis will stretched maximally, and the proximally inserted dilator measured externally to the coronal sulcus.
  Interventions: Procedure: Tumescent Stretching Measurement Technique
- Conventional Measurement technique (Active Comparator): The control group (N=12) will receive no intraoperative ICI. Following maximal corporal dilatation, cylinder length will be estimated conventionally by adding up the internally measured distal and proximal corpora to the length of the corporotomy.
  Interventions: Procedure: Tumescent Stretching Measurement Technique

INTERVENTIONS:
Procedure: Tumescent Stretching Measurement Technique — The "Tumescent Stretching Measurement Technique" (TSMT) group (N=12) will be administered an intracorporal injection (ICI) of 20 microgram Alprostadil. Hegar 7 dilator will be introduced through the corporotomy until reaching a bone stopping point. The tumescent penis will stretched maximally, and the proximally inserted dilator measured externally to the coronal sulcus.

SUMMARY:
Introducing and evaluating the accuracy of a novel method for estimating inflatable penile prosthesis cylinders length by stretching the tumesncent penis intraoperatively instead of taking proximla and distal measurement to the corporotomy

DETAILED DESCRIPTION:
Objectives:

Introducing and evaluating the accuracy of a novel method for estimating inflatable penile prosthesis cylinders length.

Methods:

24 patients undergoing a Coloplast Titan ® Touch implantation procedure will berandomly divided into two groups.

The "Tumescent Stretching Measurement Technique" (TSMT) group (N=12) will be administered an intracorporal injection (ICI) of 20 microgram Alprostadil. Hegar 7 dilator will be introduced through the corporotomy until reaching a bone stopping point. The tumescent penis will be stretched maximally, and the proximally inserted dilator measured externally to the coronal sulcus.

The control group (N=12) will receive no intraoperative ICI. Following maximal corporal dilatation, cylinder length will be estimated by adding up the internally measured distal and proximal corpora to the length of the corporotomy.

Implants are deemed correctly sized when cylinders reached the proximal third of the glans with no buckling of cylinders or floppy glans.

ELIGIBILITY:
Inclusion Criteria:

Males needing Penile implant surgery, not responding to oral pharmacological drugs for ttt of ED -

Exclusion Criteria:

Previouys penile surgery Previous implanted penile prosthesis

-

Ages: 21 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Penile Implants for Males
Enrollment: 24 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of penile implant insertions and re-insertions needed to arrive to adequate penile implant size | Intraoperative
  Number of penile implant insertions and re-insertions needed to arrive to adequate penile implant size

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR